CLINICAL TRIAL: NCT02838524
Title: Acceptable Range of Inspiratory Effort During Mechanical Ventilation
Acronym: EFFORT
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 15-369
Record Dates: First submitted 2016-07-15; First posted 2016-07-20 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Elective Cardiac Surgery
Keywords: Spontaneous Breathing Trial; Inspiratory Effort; Mechanical Ventilation; Respiratory muscle load-capacity balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Partially assisted mechanical ventilation is ideally titrated to maintain adequate inspiratory muscle activity (i.e. preventing disuse atrophy) while avoiding excessive (i.e. fatiguing) inspiratory loads. The advent of ventilator modes enabling flow and pressure assistance in proportion to patient inspiratory effort (i.e. Proportional Assist Ventilation (PAV), Neurally-Adjusted Ventilator Assist (NAVA)) permit careful titration of ventilatory support to achieve desired levels of patient inspiratory effort. However, data on the acceptable range of values for inspiratory effort and respiratory muscle load-capacity balance during mechanical ventilation are currently very limited. Such data are critical to inform a physiologically sound evidence-based approach to titrating partially-assisted ventilatory support. This study is designed to ascertain a physiologically acceptable range of inspiratory effort in mechanically ventilated patients. The study protocol includes measurements of the respiratory system during spontaneous breathing as well as evaluating the diaphragm in real-time with the use of ultrasonography. The experimental design outlined in the present study is predicated on the assumption that the range of values for inspiratory effort and load-capacity balance observed in patients who are successfully weaned from mechanical ventilation represent the safe and appropriate range of target values.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (>17) receiving invasive mechanical ventilation following elective cardiac surgery who will undergo a trial of spontaneous breathing

Exclusion Criteria:

* Pregnant women
* Decompensated cardiac insufficiency or acute coronary syndrome
* Severe COPD
* Contraindications to esophageal catheter placement, namely known esophageal varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age >17) receiving invasive mechanical ventilation following elective cardiac surgery who will undergo a trial of spontaneous breathing
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory effort generated by a patient | During 10-15 minutes of the spontaneous breathing trial

SECONDARY OUTCOMES:
Diaphragmatic thickening fraction | 15 minutes
Diaphragmatic excursion | 15 minutes
Success or failure of the spontaneous breathing trial | 15 minutes
Muscular load-capacity balance measured by the tension-time index of the respiratory muscles | 15 minutes
Airway occlusion pressure (P0.1) performed manually and as measured by the ventilator | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tobin MJ, Laghi F, Jubran A. Narrative review: ventilator-induced respiratory muscle weakness. Ann Intern Med. 2010 Aug 17;153(4):240-5. doi: 10.7326/0003-4819-153-4-201008170-00006. PMID 20713792
- [Background] Carteaux G, Mancebo J, Mercat A, Dellamonica J, Richard JC, Aguirre-Bermeo H, Kouatchet A, Beduneau G, Thille AW, Brochard L. Bedside adjustment of proportional assist ventilation to target a predefined range of respiratory effort. Crit Care Med. 2013 Sep;41(9):2125-32. doi: 10.1097/CCM.0b013e31828a42e5. PMID 23787397
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Vassilakopoulos T, Zakynthinos S, Roussos C. The tension-time index and the frequency/tidal volume ratio are the major pathophysiologic determinants of weaning failure and success. Am J Respir Crit Care Med. 1998 Aug;158(2):378-85. doi: 10.1164/ajrccm.158.2.9710084. PMID 9700110
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Lerolle N, Guerot E, Dimassi S, Zegdi R, Faisy C, Fagon JY, Diehl JL. Ultrasonographic diagnostic criterion for severe diaphragmatic dysfunction after cardiac surgery. Chest. 2009 Feb;135(2):401-407. doi: 10.1378/chest.08-1531. Epub 2008 Aug 27. PMID 18753469
- [Background] Jubran A, Tobin MJ. Pathophysiologic basis of acute respiratory distress in patients who fail a trial of weaning from mechanical ventilation. Am J Respir Crit Care Med. 1997 Mar;155(3):906-15. doi: 10.1164/ajrccm.155.3.9117025.